CLINICAL TRIAL: NCT06959446
Title: Association Between Perioperative Homocysteine and Postoperative Complications/All-Cause Mortality in Elderly Patients Undergoing Non-Cardiac Surgery
Brief Title: Perioperative Homocysteine and Postoperative Complications/All-Cause Mortality in Elderly Non-Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jingsheng Lou, Professor, Chinese PLA General Hospital
Other Study IDs: PLAGH-AOC-L07
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Elderly; Homocysteinemia; AKI - Acute Kidney Injury; Mortality; Postoperative
MeSH Terms: conditions — Homocysteinemia; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore the association between perioperative homocysteine (Hcy) levels and their pre-to-postoperative changes with postoperative complications and all-cause mortality in elderly patients undergoing non-cardiac surgery. Besides, the dynamic changes in Hcy levels may reflect metabolic shifts, highlighting their potential value in predicting adverse postoperative outcomes. These findings suggest that monitoring perioperative Hcy levels and their changes could help identify high-risk patients and inform postoperative management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized older (≥ 65 years) patients underwent non-cardiac surgery

Exclusion Criteria:

* 21227 patients without preoperative Hcy data
* 957 patients undergoing neurosurgery
* 3 patients call off the surgery for reasons
* 164 patients with chronic kidney disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: An observational study using data from the First Medical Center of Chinese PLA General Hospital, an electronic medical record-based data set of 12,955 older patients (≥ 65 years) who had surgery between January 2014 to August 2019
Sampling Method: Non-Probability Sample
Enrollment: 12955 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury (AKI) | January 2014 - August 2019

SECONDARY OUTCOMES:
mortality | January 2014 - August 2020